CLINICAL TRIAL: NCT02053103
Title: A 6-Week Phase 2a Randomized, Double-Blind, Placebo-Controlled Study To Assess Safety, Tolerability And Pharmacodynamics Of Oral PF-05175157 In Adult Subjects With Type 2 Diabetes Mellitus Inadequately Controlled On Metformin
Brief Title: A 6-Week Study To Determine The Safety And Effect Of An Investigational Drug On Adults With Type 2 Diabetes Mellitus Taking Metformin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: On 25April2014, study was terminated before any dosing due to an AE of safety concern that occurred in protocol B1731003 with the same drug.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1731002
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-05175157 (Experimental)
  Interventions: Drug: PF-05175157
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05175157 — Tablet, 200 mg, twice daily, 6 weeks
  Arms: PF-05175157
Drug: Placebo — Tablet, 0 mg, twice daily, 6 weeks
  Arms: Placebo

SUMMARY:
A Phase 2a study to evaluate the effects of an investigational compound administered at 200 mg, twice daily (BID), for 6 weeks in adult subjects with Type 2 Diabetes Mellitus (T2DM) on metformin background therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus and treated with metformin at a dose greater than or equal to 1000 mg for at least 3 months
* Hemoglobin A1c of 7-10% at screening.
* Body Mass Index of at least 25 kg/m2.

Exclusion Criteria:

* Compliant with study drug administration during the run-in period and throughout the trial.
* Patients with fasting triglycerides greater than 500 mg/dL at screening.
* History of certain diabetic complications or cardiac problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Weighted Mean Daily Glucose (WMDG) when compared to placebo | Baseline, Day 42

SECONDARY OUTCOMES:
Change from baseline in Weighted Mean Daily Glucose (WMDG) when compared to placebo | Weeks 0 and 4
Change from baseline in fasting plasma glucose | Weeks 0, 2, 4 and 6
Change from baseline in Glycosylated Hemoglobin (HbA1c) | Weeks 0, 4 and 6
Change from baseline in fasting total cholesterol | Weeks 0, 4 and 6
Change from baseline in glucose AUC(0-5) during mixed meal tolerance test (MMTT) | Weeks 0, 4 and 6
Change from baseline in insulin AUC(0-5) during mixed meal tolerance test (MMTT) | Weeks 0, 4 and 6
Change from baseline in ratio of AUC (0-5) C-peptide to AUC(0-5) glucose during the MMTT | Weeks 0, 4 and 6
Change from baseline in ratio of AUC(0-5) insulin to AUC(0-5) glucose during the MMTT | Weeks 0, 4 and 6
Change from baseline in homeostatic model assessment for insulin resistance (HOMA IR) | Weeks 0, 4 and 6
Change from baseline in homeostatic model assessment for β-cell function (HOMA B) | Weeks 0, 4 and 6
Plasma concentrations for PF-05175157 | Weeks 2, 4 and 6
Percent change from baseline in body weight | Weeks 0, 4 and 6
Change from baseline in low density lipoprotein cholesterol (LDL-C) | Weeks 0, 4 and 6
Change from baseline in high density lipoprotein cholesterol (HDL-C) | Weeks 0, 4 and 6
Change from baseline in triglycerides | Weeks 0, 4 and 6
Change from baseline in non-HDL cholesterol | Weeks 0, 4 and 6
Change from baseline in very low density lipoprotein (VLDL) | Weeks 0, 4 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Orlando, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1731002&StudyName=A%206-Week%20Study%20To%20Determine%20The%20Safety%20And%20Effect%20Of%20An%20Investigational%20Drug%20On%20Adults%20With%20Type%202%20Diabetes%20Mellitus%20Taking%20Metformi